CLINICAL TRIAL: NCT03370718
Title: A Phase II Study to Evaluate the Effects of Cabozantinib in Patients With Unresectable/Metastatic Adrenocortical Carcinoma
Brief Title: Cabozantinib in Treating Patients With Locally Advanced or Metastatic Unresectable Adrenocortical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0741; NCI-2018-00973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0741 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-12-08; First posted 2017-12-12 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Carcinoma in the Adrenal Cortex; Stage III Adrenal Cortex Carcinoma AJCC v8; Stage IV Adrenal Cortex Carcinoma AJCC v8; Unresectable Adrenal Cortex Carcinoma
MeSH Terms: conditions — Adrenal Cortex Neoplasms | interventions — cabozantinib; Pharmacogenomic Testing; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib) (Experimental): Patients receive cabozantinib PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Other: Pharmacogenomic Study; Other: Pharmacokinetic Study

INTERVENTIONS:
Drug: Cabozantinib — Given PO
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase II trial studies how well cabozantinib works in treating patients with adrenal cortex cancer that has spread to nearby tissue, lymph nodes (locally advanced), or other places in the body (metastatic), and cannot be removed by surgery (unresectable). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate progression free survival at 4 months.

SECONDARY OBJECTIVES:

I. Best overall response rate. II. Overall survival (OS). III. Toxicity assessment by the Common Terminology Criteria for Adverse Events (CTCAE) version (V)4.0.

EXPLORATORY OBJECTIVES:

I. Pharmacokinetics and cabozantinib serum levels to assess correlation with response to therapy.

II. Steroid hormone biomarkers as markers of disease response. III. Study the effect of cabozantinib on immune markers by obtaining optional biopsy and blood samples collections at baseline, during therapy and at time of progression.

IV. Pharmacogenomics of drug disposition gene variants that potentially influence cabozantinib pharmacokinetics (PK).

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30-37 days.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adrenocortical carcinoma (ACC) based on either: i). Weiss Score of >= 3 in patients who had earlier surgical resection OR ii). biopsy results compatible with ACC in the context of clinical setting highly suggestive of ACC (adrenal mass > 4 cm invading surrounding organs or associated with distant metastases).
* Locally advanced or metastatic disease not amenable to surgery with curative intent with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the investigator based on an assessment of all known disease sites by computerized tomography (CT) scan or magnetic resonance imaging (MRI) of chest/abdomen/pelvis within 28 days before the first dose of cabozantinib. In patients with intravenous (IV) contrast allergy or borderline renal function, CT without IV contrast or 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) CT may be used as clinically indicated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Recovery to baseline or =< grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless adverse events (AEs) are clinically nonsignificant and/or stable on supportive therapy.
* Life expectancy of at least 3 months.
* Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support (obtained within 28 days prior to the first dose of cabozantinib).
* Platelets >= 100,000/mm^3 (obtained within 28 days prior to the first dose of cabozantinib).
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to the first dose of cabozantinib).
* Bilirubin =< 1.5 x the upper limit of normal (ULN). For subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL (obtained within 28 days prior to the first dose of cabozantinib).
* Serum albumin >= 2.8 g/dl (obtained within 28 days prior to the first dose of cabozantinib).
* Serum creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 50 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used (obtained within 28 days prior to the first dose of cabozantinib).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN (obtained within 28 days prior to the first dose of cabozantinib).
* Lipase =< 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis (obtained within 28 days prior to the first dose of cabozantinib).
* Urine protein/creatinine ratio (UPCR) =< 1 (obtained within 28 days prior to the first dose of cabozantinib).
* Serum phosphorus >= 2.5 mg/dl (obtained within 28 days prior to the first dose of cabozantinib).
* Calcium >= 8 mg/dL (obtained within 28 days prior to the first dose of cabozantinib).
* Magnesium >= 1.2 mg/dL (obtained within 28 days prior to the first dose of cabozantinib).
* Potassium >= 3.0 meq/L (obtained within 28 days prior to the first dose of cabozantinib).
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active patients (men and women) must agree to use medically accepted barrier methods of contraception (e.g. male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All sexually active subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).
* Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea >= 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible reason.

Exclusion Criteria:

* Received cytotoxic chemotherapy, radiation therapy, or targeted therapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 28 days of study enrollment.
* For patients who received mitotane within 6 months of consenting, mitotane should have been stopped at least 28 days prior to study enrollment AND to have mitotane serum level of < 2 mg/L.
* Prior treatment with cabozantinib or other cMET inhibitors.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment.
* The subject has not recovered to baseline or CTCAE =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs.
* Prothrombin time (PT)/ international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 28 days before the first dose of study treatment.
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors), platelet inhibitors (e.g., clopidogrel) or therapeutic doses of low molecular weight heparins (LMWH). Low dose aspirin for cardioprotection (per local applicable guidelines) and low-dose LMWH are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects who are on a stable dose of LMWH for at least 6 weeks before the first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Severe and uncontrolled Cushing syndrome despite medical management (e.g., systolic blood pressure > 160 mmHg or hyperglycemia with fasting glucose above 300 mg/dL).
* The use of strong CYP3A4 inhibitor (with the exception of ketoconazole).
* The subject has experienced any of the following: a. clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment; b. hemoptysis >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment; c. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment. Tumor invading any major blood vessel at the time of study enrollment.
* Evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib, or the subject with radiographic evidence of cavitating pulmonary lesion(s); or subjects with tumor invading or encasing any major blood vessels.
* Uncontrolled, significant concurrent or recent illness including, but not limited to, the following conditions: a. Cardiovascular disorders including i. congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening ii. concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment iii. any history of congenital long QT syndrome or iv. any of the following within 6 months before the first dose of study treatment: unstable angina pectoris, clinically-significant cardiac arrhythmias, stroke (including transient ischemic attack [TIA], or other ischemic event) within 90 days of the first dose of study treatment, myocardial infarction, clinically significant thromboembolic event within 42 days of randomization requiring therapeutic anticoagulation.
* (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study) b. gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including: i. any of the following within 28 days before the first dose of study treatment: intra-abdominal tumor/metastases invading GI mucosa, active peptic ulcer disease; patients must be completely recovered, inflammatory bowel disease (including ulcerative colitis and Crohn's disease), acute pancreatitis, pancreatic duct or common bile duct obstruction, acute diverticulitis, acute cholecystitis, symptomatic cholangitis or recent appendicitis within 1 month of first dose of cabozantinib; patients must be completely recovered from these conditions, clinically significant malabsorption syndrome, c. endocrine disorders, uncontrolled Cushing syndrome despite of adequate medical therapy.
* Any of the following within 6 months before the first dose of study treatment: abdominal fistula, gastrointestinal perforation, bowel obstruction or gastric outlet obstruction, intra-abdominal abscess. Note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment. Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 90 days before the first dose of study therapy.
* Other clinically significant disorders such as: i. active infection requiring systemic antibiotic treatment within 14 days before the first dose of study treatment ii. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment iii. history of organ transplant iv. concurrent uncompensated hypothyroidism or thyroid dysfunction (thyroid-stimulating hormone [TSH] above 10) within 28 days before the first dose of study treatment v. major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Unable to swallow tablets.
* A corrected QT interval calculated by the Fridericia formula (QTcF) > 500 milliseconds within 28 days before first dose of study treatment.
* Pregnant or breastfeeding.
* A previously identified allergy or hypersensitivity to components of the study treatment formulation.
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* Evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment except for breast ductal carcinoma-in situ, cured non-melanoma skin cancer, or cured in situ cervical carcinoma.
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality which, in the judgment of the investigator, would have made the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouhammed A Habra, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Campbell MT, Balderrama-Brondani V, Jimenez C, Tamsen G, Marcal LP, Varghese J, Shah AY, Long JP, Zhang M, Ochieng J, Haymaker C, Habra MA. Cabozantinib monotherapy for advanced adrenocortical carcinoma: a single-arm, phase 2 trial. Lancet Oncol. 2024 May;25(5):649-657. doi: 10.1016/S1470-2045(24)00095-0. Epub 2024 Apr 9. PMID 38608694
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study assessed 28 patients for eligibility, 18 started treatment, and at present none remained on therapy.
Groups:
- Cabozantinib: Patients with advanced adrenocortical carcinoma meeting inclusion and exclusion criteria
Period: Overall Study
Arm/Group | Cabozantinib
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 55.5 [46.3 to 64.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria
Description: PFS rates will be monitored simultaneously using the Bayesian approach of Thall, Simon, Esty as extended by Thall and Sung. PFS is defined as no disease progression or death within the first 4 months of the proposed treatment.
Time Frame: At 4 months
Measure: Number (95% Confidence Interval); unit: precentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 18
precentage of participants | 72.2 [46.5 to 90.3]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years and 3 months
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=18)
Abdominal pain (Gastrointestinal disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 11
Anemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3
Belching (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 6
Bruising (Injury, poisoning and procedural complications) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cortisol increase (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 7
Decreased Chloride (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema/Rash (Investigations) | 5
Extremity pain (Musculoskeletal and connective tissue disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Free T4 alteration (Blood and lymphatic system disorders) | 2
Gait disturbance (General disorders) | 1
GGT increased (Investigations) | 2
Gingival pain (Infections and infestations) | 1
Hair color changing (Skin and subcutaneous tissue disorders) | 4
Hair loss (Skin and subcutaneous tissue disorders) | 1
Hand pain/ joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 5
Heat intolerance (General disorders) | 2
Hematemesis (Blood and lymphatic system disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Hypothyroidism (Endocrine disorders) | 3
Increased amylase (Investigations) | 7
Increased BUN (Investigations) | 1
Increased calluses on feet (Skin and subcutaneous tissue disorders) | 2
Increased GGT (Investigations) | 7
Increased Globulin (Investigations) | 1
Increased LDH (Blood and lymphatic system disorders) | 7
Increased PT (Blood and lymphatic system disorders) | 1
Increased PTT (Investigations) | 2
Increased skin sensitivity (Investigations) | 1
Increased T4 (Endocrine disorders) | 1
Increased Total Protein (Investigations) | 1
Increased TSH (Endocrine disorders) | 8
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 4
Intracranial hemorrhage (Nervous system disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Lightheadedness (Investigations) | 2
Lipase increased (Investigations) | 8
Loss of Peripheral vision (Eye disorders) | 1
Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mucositis oral (Gastrointestinal disorders) | 6
Muscle cramps (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discharge (General disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Odynophagia (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pallor (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Pancreatitis (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 3
Peeling and Dry blistering (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia bibasilar (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 9
Radiculitis (Nervous system disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 5
Skin infection (Skin and subcutaneous tissue disorders) | 1
Slow growth of hair (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Soreness on sole of feet (Musculoskeletal and connective tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Thyrotoxicosis (Endocrine disorders) | 1
Total Protein decreased (Blood and lymphatic system disorders) | 1
Tremor (Nervous system disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteral obstruction (Renal and urinary disorders) | 1
Urinary hesitancy (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Voice change (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Weight gain (Investigations) | 1
Weight loss (Investigations) | 12
White blood cell decreased (Investigations) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03370718/Prot_SAP_000.pdf